CLINICAL TRIAL: NCT05123690
Title: Neurofeedback for Post-Traumatic Stress Disorder (N-PTSD). A Randomized Trial of Neurofeedback.
Brief Title: Neurofeedback for Post-Traumatic Stress Disorder
Acronym: ViN-PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steinn Steingrimsson (Other)
Responsible Party: Sponsor-Investigator, Steinn Steingrimsson, Principal investigator & clinical associate professor, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNF001
Record Dates: First submitted 2021-09-20; First posted 2021-11-17 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Post-traumatic Stress Disorder
Keywords: Neurofeedback; Electroencephalogram (EEG)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neurofeedback; Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Allocation is to one of two arms
Masking Description: Statistical analysis will be done seperately
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback (Experimental): 24 sessions of ca 45 minutes neurofeedback using alpha-theta protocol.
  Interventions: Device: Neurofeedback
- Waiting list (No Intervention): Those assigned to waiting list will be able to pick one of the two interventions at the end of the study.

INTERVENTIONS:
Device: Neurofeedback — A device that assists in training patients in relaxing.
  Other Names: EEG assisted neurofeedback; Biofeedback
  Arms: Neurofeedback

SUMMARY:
A two-arm randomized pilot of standard neurofeedback and a waiting list for patients with treatment resistent PTSD.

DETAILED DESCRIPTION:
This study will be a randomized-controlled pilot and in a later study virtual reality based neurofeedback will be tested. In this study 30 subjects will be randomised into one of two arms of the study. Treatment as usual (TAU) entails both psychotherapy, medication and other interventions.

1. TAU + Neurofeedback using a PC-screen (experimental group)
2. TAU as a waiting list (control group) - the participants in the control group will be offered to choose one of the two experimental treatments at the end of the trial.

The 30 participants will be randomized to one arm of the study (15 participants per group). The subjects will be recruited from Psychiatric Outpatient Care at Sahlgrenska University Hospital, Crisis and Trauma Center Gothenburg and Psychiatric Care Center in Tranås, Jönköping.

Participants in the experimental group will have 24 sessions in total, (twice a week. 12 week period) with a trained neurofeedback specialist or trained neurofeedback physician. Before session 1 and after session 24, a clinician will fill in the clinical scales and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* CAPS Cutoff >44
* Stable psychopharmacological treatment (stable dose, no planned changes during the course of the trial)
* AUDIT cut off <16
* DUDIT cut off <8
* Already undergone at least one treatment with psychotherapy and/or pharmacological treatment for a minimum of 6 months.
* 18 years or older

Exclusion Criteria:

* Diagnosis of traumatic brain injury (TBI) affecting capability to give informed consent
* Ongoing traumatic exposure (such as domestic violence)
* Balance problems
* Active suicide risk or life-threatening self-harm
* A diagnosis of schizophrenia or psychotic disorder
* Ongoing compulsory care
* If the patient changes dose or medication strategy during the trial.
* If the neurofeedback treatment is identified as a primary reason for worsening of participant's well being.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Through study completion, an average of 3 months
  An interview based scale of symptoms of PTSD

SECONDARY OUTCOMES:
Impact of Event Scale - Revised (IES-R) | Through study completion, an average of 3 months
  IES-R is a self-assessment scale that measures the degree to which one has been affected by post-traumatic stress reactions during the last 7 days.
Impact of Event Scale - Revised (IES-R) | 4 weeks after finished intervention for the two intervention arms.
  IES-R is a self-assessment scale that measures the degree to which one has been affected by post-traumatic stress reactions during the last 7 days.
Visual Analogue Scale for Wellbeing (VAS-W) | Before and after each session 1-24 for the two intervention arms.
  The measurement is a 10 point scale ranging from 1-10 with a visual representation (a sad face at 1 and happy face at 10) asking "How are you feeling right now".
Insomnia Severity Index (ISI) | Through study completion, an average of 3 months
  The scale consists of 7 items where participants can score their sleep quality and frequency on a scale from 0-4. 0 being no problems while 4 meaning significant problems. The score ranges from 0-28.
Insomnia Severity Index (ISI) | 4 weeks after finished intervention for the two intervention arms.
  The scale consists of 7 items where participants can score their sleep quality and frequency on a scale from 0-4. 0 being no problems while 4 meaning significant problems. The score ranges from 0-28.
Wisconsin Card Sorting Test (WCST) | Through study completion, an average of 3 months
  A cognitive test measuring attention, vigilance and memory.
Wisconsin Card Sorting Test (WCST) | 4 weeks after finished intervention, an average of 4 months
  A cognitive test measuring attention, vigilance and memory.
Clinician Administered PTSD Scale (CAPS) | For those that have finished the intervention CAPS at one month post treatment
  An interview based scale of symptoms of PTSD

CONTACTS AND LOCATIONS:
Overall Officials: Steinn Steingrimsson, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No
This will be discussed if the occasion arises in order to follow GDPR and ethical rules.